CLINICAL TRIAL: NCT02575040
Title: Efficacy of Fecal Microbiota Transplantation for Refractory Inflammatory Bowel Disease
Brief Title: Efficacy of Fecal Microbiota Transplantation for Inflammatory Bowel Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Hakan Demirci, doctor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMMA-Fecal Tx-1
Record Dates: First submitted 2015-10-06; First posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Ulcerative Colitis; Crohn Disease; Constipation (Excl Faecal Impaction)
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Constipation | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fecal microbiota transplantation (Other): Fecal microbiota transplantation only
  Interventions: Biological: Fecal microbiota transplantation

INTERVENTIONS:
Biological: Fecal microbiota transplantation — Fecal microbiota transplantation to patients with ulcerative colitis and Crohn disease

SUMMARY:
The gut microbiota is determined to constitute a "microbial organ" which has pivotal roles in the intestinal diseases and body's metabolism. Evidence from animal and human studies strongly supports the link between intestinal bacteria flora and inflammatory bowel diseases. Lots of studies showed its efficacy in treatment of severe Clostridium difficile colitis. Corticosteroid dependence in patients with ulcerative colitis (UC) and Crohn's disease (CD) is an important clinical problem and maintenance of steroid-free remission is a key treatment goal. Early studies using fecal microbiota transplantation (FMT) for Ulcerative Colitis (UC) and Crohn's diseases have also met with success. This is an first step into investigating the potential efficacy of standardized FMT through terminal ileum for UC and CD, the investigators propose to determine the efficiency and safety of FMT in a series of 80 patients with moderate to severe UC and CD.

DETAILED DESCRIPTION:
Intestinal microbiota have a major role in disease pathogenesis, either in a form of a "permissive" role or as a direct pathogenic cause.

Clostridium difficile colitis; irritable bowel syndrome (IBS) and inflammatory bowel disease (IBD) have all been connected to a disturbance in the equilibrium of intestinal microbiome. The cause of IBD in unknown but evidence is getting that immense immune reaction of intestinal immune system to microflora combined with a genetic predisposition are responsible for the chronic inflammation.

Fecal microbial treatment (FMT) is a treatment that utilizes the microbiota of a healthy intestine as a probiotic preparation. The fecal material of a healthy individual is fluidized and that inserted into the intestinal tract of a sick individual, assuming that the healthy flora will colonize and cure the intestine. Previous work had shown success in fecal transplantation as a treatment for clostridium difficile colitis. There are also reports of the efficacy of this treatment for inflammatory bowel disease but currently the numbers are small. 41 cases were reported , In some the FMT was inserted through a nasogastric tube directly to the duodenum, in some be colonoscopy and in some by an enema. A significant clinical improvement was reported in 19 of 25 patients. 13 of 17 stopped IBD treatment , 15 of 24 entered full clinical remission. In all 15 patients treated for infection the treatment was successful. No sever adverse effects were reported, Fever was developed in 8 cases and in one case there was exacerbation of colitis after treatment.

Primary aim: To investigate whether use of FMT will bring improvement of at least 2 points in partial mayo score in ulcerative colitis patients, or 75 points in CDAI of patients with Crohn's colitis. One month after FMT.

Improvement will be defined as:

For Ulcerative colitis: a decrease of at least 2 points in the partial mayo score, and a decrease of at least 1 point in endoscopic Mayo score.

For Crohn's disease: A decrease of at least 70 points in Crohn's disease activity index (CDAI).

80 patients aged >18 years, with histological and endoscopic diagnosis of ulcerative colitis (UC) or CD who did not respond to either thiopurines or tumor necrosis factor (TNF) inhibitors.

Flare will be defined as partial mayo score higher then 3, with either C reactive protein (CRP) higher than 6 or endoscopic mayo score >1 in ulcerative colitis and CDAI higher them 220 and CRP higher than 6 in Crohn's colitis.

Stool will be donated by the patients choice either from a relative, preferably a partner to minimize possible transference of an infective agent, alternatively samples will be ordered from "open biom".

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Inflammatory bowel disease diagnosed at least 6 months ago
* Failure of either one immunomodulator of at least 3 months duration, or TNF inhibitor full induction treatment, or corticosteroids, or intolerance to either of these drugs.
* Currently active disease, partial Mayo score ≥4 for ulcerative colitis, or CDAI ≥200 for CD.
* negative HIV , Human T-cell leukemia virus I/II, negative stool culture, Negative C diff toxin, negative Cytomegalovirus

Exclusion Criteria:

* No informed consent
* Non active inflammatory bowel disease.
* Active infection in either the donor or the recipient,
* Response to biological agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Patients with worsened disease | one year
  Number of patients with worsened disease. Increase in Montreal score S1, S2 and S3.
Adverse events | one year
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Uygun, Prof, Principal Investigator — Gulhane Military Medical Academy, Department of Gastroenterology
Locations (1):
- Gulhane Military Medical Academy, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Cui B, Li P, Xu L, Zhao Y, Wang H, Peng Z, Xu H, Xiang J, He Z, Zhang T, Nie Y, Wu K, Fan D, Ji G, Zhang F. Step-up fecal microbiota transplantation strategy: a pilot study for steroid-dependent ulcerative colitis. J Transl Med. 2015 Sep 12;13:298. doi: 10.1186/s12967-015-0646-2. PMID 26363929
- [Result] Wei Y, Zhu W, Gong J, Guo D, Gu L, Li N, Li J. Fecal Microbiota Transplantation Improves the Quality of Life in Patients with Inflammatory Bowel Disease. Gastroenterol Res Pract. 2015;2015:517597. doi: 10.1155/2015/517597. Epub 2015 Jun 4. PMID 26146498
- [Result] Rossen NG, MacDonald JK, de Vries EM, D'Haens GR, de Vos WM, Zoetendal EG, Ponsioen CY. Fecal microbiota transplantation as novel therapy in gastroenterology: A systematic review. World J Gastroenterol. 2015 May 7;21(17):5359-71. doi: 10.3748/wjg.v21.i17.5359. PMID 25954111
- [Derived] Uygun A, Ozturk K, Demirci H, Oger C, Avci IY, Turker T, Gulsen M. Fecal microbiota transplantation is a rescue treatment modality for refractory ulcerative colitis. Medicine (Baltimore). 2017 Apr;96(16):e6479. doi: 10.1097/MD.0000000000006479. PMID 28422836